CLINICAL TRIAL: NCT02945683
Title: Randomized Controlled Trial to Evaluate the Beneficial Effects of a Probiotic Food Supplement in Children With Atopic Dermatitis
Brief Title: Effects of Lactobacillus Reuteri Plus Vitamin D3 in Children With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noos S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ATOPIA_D3
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis, probiotics, vitamin D3, L. reuteri
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reuterin D3 (Active Comparator): Patients should take 10 drops once a day during meals for 3 months
  Interventions: Dietary Supplement: Reuterin D3
- Placebo (Placebo Comparator): Patients should take 10 drops once a day during meals for 3 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Reuterin D3 — Lactobacillus reuteri DSM 17938 (10E8 CFU in 5 drops), Vitamin D3 (400 IU in 5 drops), sunflower oil, medium chain triglycerides, silicon dioxide
  Arms: Reuterin D3
Dietary Supplement: Placebo — sunflower oil, medium chain triglycerides, silicon dioxide
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate in a randomized, double-blinded, controlled trial, whether a new food supplement containing Lactobacillus reuteri DSM 17938 and vitamin D3 (Reuterin® D3) may improve the SCORAD in pediatric patients with mild to moderate atopic dermatitis

DETAILED DESCRIPTION:
Recent evidence suggests that childhood allergy development can be linked to an imbalance of the intestinal microbiota. The probiotic bacteria, which contribute to the balance of the intestinal microflora, may play a key role in the modulation of the immune response, looking as a potential resource in the prevention or treatment of allergic disorders.

In this study the investigators will recruit pediatric patients with atopic dermatitis of mild-to-moderate degree, for which the standard treatment consists in using an emollient cream and topical steroids in case of exacerbation.

The investigators assume that participants can receive significant benefits from the addition to their standard treatment of a food supplement containing L. reuteri DSM 17938 and vitamin D3, which, thanks to their beneficial effects on intestinal microbiota and on modulation of the immune response, may compensate for the inadequate capacity of these patients to produce antimicrobial peptides in response to cutaneous aggressions, improving, therefore, the severity of the disease.

88 children of both sexes, between 1 and 4 years old, with a SCORAD of 25-50 will be selected as a part of routine outpatient visits at the Pediatric Allergy Department of the University Hospital of Verona.

The study product (active or placebo) will be administered for 3 months, with a follow-up period of further 3 months. From all participants, at time 0 and after 3 months, blood and stool samples will be collected for the analysis of vitamin D and cathelicidin levels and for the analysis of microflora respectively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of atopic dermatitis of mild to moderate grade (SCORAD 25-50)
* signature of the informed consent from both parents or a legal representative

Exclusion Criteria:

* presence of autoimmune diseases, immunodeficiency, inflammatory bowel diseases, cystic fibrosis, metabolic diseases
* use of immunosuppressive drugs and/or systemic corticosteroids in the previous 2 months
* use of antibiotics in the last 4 weeks
* use of probiotics and/or prebiotics in the last 2 weeks
* use of vitamin D in the last 4 weeks
* participation in other clinical trials

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
SCORAD improvement | 3 months
  Improvement of the SCORAD compared to baseline

SECONDARY OUTCOMES:
Vitamin D levels increase | 3 months
  Increase of the levels of Vit. D compared to baseline
LL-37 levels increase | 3 months
  Increase of the levels of cathelicidin compared to baseline
Changes in the fecal microflora | 3 months
  Changes in the fecal microflora compared to baseline
QoL improvement | 3 months
  Improvement of the child's quality of life

OTHER OUTCOMES:
Food Frequency Questionnaire | 3 months
  Evaluation of the child's eating habits

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Boner, Professor, Principal Investigator — Policlinico G.B. Rossi, Head of the Pediatric Department
Locations (1):
- Policlinico G.B. Rossi, Verona, Italy

IPD SHARING:
Plan to Share IPD: No